CLINICAL TRIAL: NCT00317057
Title: Outpatient Management of Patients With Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: KA05756
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; Outpatient management; nurse-lead patient education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Patient Education as Topic; Disease Management

INTERVENTIONS:
Procedure: Patient education and disease management

SUMMARY:
Patients admitted to the hospital with chronic obstructive pulmonary disease are evaluated with regard to early follow-up by a specialized nurse in the home after discharge.

DETAILED DESCRIPTION:
Patients admitted to Department of Internal Medicine M, Glostrup University hospital, with Chronic Obstructive Pulmonary Disease (COPD) are evaluated with regard to early follow-up by a specialized nurse in the home after discharge. Eligible patients receive education about disease management. The intervention is evaluated by comparing the number of readmissions for COPD and the duration of admissions during the study period to the the period prior to the implementation of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Admission for chronic obstructive pulmonary disease

Exclusion Criteria:

* Other severe acute or chronic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2006-04; Study Completion 2007-01

PRIMARY OUTCOMES:
the number of readmissions for chronic obstructive pulmonary disease

SECONDARY OUTCOMES:
the duration of admissions for chronic obstructive pulmonary disease

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Vest, MD, Principal Investigator — Glostrup University Hospital, Copenhagen; Allan Linneberg, MD, PhD, Study Chair — Glostrup University Hospital, Copenhagen
Locations (1):
- Department of Internal Medicine, Glostrup University Hospital, Copenhagen, Glostrup, Denmark